CLINICAL TRIAL: NCT03003793
Title: Insulin Sensitivity in Patients With Atopic Dermatitis
Acronym: AD-IF
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD PhD, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-15010198
Record Dates: First submitted 2016-03-01; First posted 2016-12-28 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis/Eczema; Type 2 Diabetes
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Healthy control subjects
  Interventions: Diagnostic Test: Hyperinsulinemic euglycemic clamp
- Atopic dermatitis/eczema group: Patients with atopic dermatitis
  Interventions: Diagnostic Test: Hyperinsulinemic euglycemic clamp

INTERVENTIONS:
Diagnostic Test: Hyperinsulinemic euglycemic clamp — Hyperinsulinemic euglycemic clamp to detect insulin sensitivity

SUMMARY:
The incidence of atopic dermatitis and type 2 diabetes, respectively, has increased over many years. Novel research shows an association between the two conditions. While this relationship at least in theory can be explained by lifestyle factors, there is reason to believe that other pathophysiological mechanisms are involved. Hence, our hypothesis is that patients with atopic dermatitis are insulin resistant due to their chronic inflammatory state. Insulin resistance might play an unknown part in the increased frequency of type 2 diabetes among patients with atopic dermatitis. In the present project, the investigators aim to measure insulin sensitivity by means of the 'golden standard' hyperinsulinaemic euglycaemic clamp in patients suffering from atopic dermatitis compared to a healthy control group (matched case-control study). The project is a close collaboration between The Department of Dermatology and Allergy and Center for Diabetes Research at Gentofte Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe atopic dermatitis for at least 5 years
* BMI < 30 kg/m2
* HbA1c < 42 mmol/mol

Exclusion Criteria:

* Diabetes
* Prediabetes
* First-degree relatives with diabetes
* Chronic inflammatory diseases other than atopic dermatitis and asthma
* Pregnancy
* Breast-feeding
* Daily intake of medications that are known to influence the glucose metabolism are not allowed one month before the study (e.g. asthma medicines and hormonal contraception).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with atopic dermatitis are recruited from Department of Dermatology and Allergology at Gentofte Hospital.
  Control subjects are recruited from the Danish recruitment site "www.forsoegsperson.dk".
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — University Hospital, Gentofte; Jacob P Thyssen, MD,PhD,DMSc, Study Director — University Hospital, Gentofte
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Healthy control subjects Hyperinsulinemic euglycemic clamp
- Atopic Dermatitis/Eczema Group: Patients with atopic dermatitis Hyperinsulinemic euglycemic clamp
Period: Overall Study
Arm/Group | Control Group | Atopic Dermatitis/Eczema Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Atopic Dermatitis/Eczema Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (3) | 33 (3) | 33 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Denmark | 16 | 16 | 32
Atopic dermatitis duration [Mean (Standard Deviation); unit: years] | NA (NA) — No atopic dermaitits in this group | 28 (3) | NA (NA) — Only atopic dermaitits in one of the groups.
Body master index [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (1) | 24.5 (1) | 24.5 (1)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Difference Between Patients With Atopic Dermatitis and Controls
Description: The outcome is determined by measuring the glucose necessary to maintain euglycaemia during increased insulin levels generated by continuous insulin infusion (measured as the M-value: the rate of glucose infused is equal to the rate of whole-body glucose disposal or metabolizable glucose (M) and reflects the amount of exogenous glucose necessary to fully compensate for the hyperinsulinemia)
Time Frame: Baseline, plasma glucose every 5 minutes, insulin/C-peptide, glucagon every 10-15 minutes throughout a 3 hour hyperinsulinaemic euglycaemic clamp
Measure: Mean (Standard Deviation); unit: mg glucose/kg body mass/minute
Arm/Group | Control Group | Atopic Dermatitis/Eczema Group
Number analyzed (Participants) | 16 | 16
mg glucose/kg body mass/minute | 9.8 (0.8) | 9.2 (0.6)

ADVERSE EVENTS:
Arm/Group | Control Group | Atopic Dermatitis/Eczema Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes